CLINICAL TRIAL: NCT05100706
Title: Continuous Adductor Canal Block in Outpatient Total Knee Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other)
Responsible Party: Principal Investigator, Hermann dos Santos Fernandes, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-0041-A
Record Dates: First submitted 2021-09-28; First posted 2021-10-29 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Knee Arthroplasty, Total; Anesthesia, Regional; Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled prospective trial, blinded for patient and evaluator, in patients undergoing outpatient primary TKA at Sinai Health.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized to one of the two groups using a computer-generated random numbers table. The randomization will be done before the beginning of the study and will define which study number is going to be managed as interventional group (continuous adductor canal block - CACB) or control group (sham continuous adductor canal block - ShACB). Each patient will receive a study number following the order of their entrance on the study. The elastomeric pumps to be used connected to the catheter will be previously prepared by hospital pharmacy, accordingly to the randomization made and the subject study number, with no identification of the content (NaCl 0.9% or Ropivacaine 0.2%). Hospital pharmacy will not be blinded for which study number and elastomeric pump will be linked to the study group. Research coordinator, professional who performs the adductor canal catheter insertion and researcher who collects the data will be blinded to which group each patient was randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous adductor canal block (CACB) (Experimental): Will receive an infusion of 0.2% ropivacaine 5mL/h through adductor canal catheter.
  Interventions: Drug: Continuous adductor canal block (CACB)
- Sham continuous adductor canal block (ShACB). (Placebo Comparator): Will receive an infusion of NaCl 0.9% 5mL/h through adductor canal catheter.
  Interventions: Drug: Sham continuous adductor canal block (ShACB).

INTERVENTIONS:
Drug: Continuous adductor canal block (CACB) — Ropivacaine 0.2% infusion through adductor canal catheter
  Arms: Continuous adductor canal block (CACB)
Drug: Sham continuous adductor canal block (ShACB). — NaCl 0.9% infusion through adductor canal catheter
  Arms: Sham continuous adductor canal block (ShACB).

SUMMARY:
Total knee arthroplasty (TKA) is a frequent performed surgery. Many institutions are implementing outpatient programs for this surgery and adequate pain management is an important feature. Analgesic duration of single shot nerve blocks is limited to no more than 24h. Conversely, the use of continuous nerve block (CNB) through a perineural catheter and infusion of local anesthetic may increase duration of analgesia and provide better outcomes. The purpose of this study is to evaluate effectiveness and safety of using CNB in patients undergoing primary TKA, and its effects on patients' quality of recovery. We hypothesize that continuous adductor canal block would lead to a better quality of recovery in patients undergoing primary TKA.

DETAILED DESCRIPTION:
Objectives: Evaluate effectiveness and safety of using continuous adductor canal block (CACB) in patients undergoing primary total knee arthroplasty (TKA), in comparison to single shot adductor canal block (SACB). Primary objective is assess the quality of recovery of those patients (using the 15-item quality of recovery scale - QoR-15) at predetermined time points postoperatively. Secondary objectives are to evaluate postoperative pain scores, postoperative use of opioid, postoperative functional status, complications relating to the perineural catheter.

Hypothesis: Continuous adductor canal block would lead to a better quality of recovery in patients undergoing primary TKA.

Methods: Randomized controlled prospective trial, blinded for patient and evaluator, in patients undergoing primary TKA at Sinai Health. After Hospital's Ethics in Research Board approval, the recruitment will begin. Patients will be assessed about their eligibility for participating and after plain clear information about the study interventions they will or will not authorize their inclusion and data collection, through the signature of a written consent. The subjects will have their surgeries booked in advance and they will be submitted to the pre anesthesia consult at the Pre Admission Unit a few days before the surgery. The study proposal will be explained to the patients in that occasion. They will receive a booklet with information about the study and the Consent Form that they will bring home with them. They will have the time between the pre anesthesia assessment and the surgery (at least two days) to review and consent to the study. Patients will be randomized to one of the two groups using a computer-generated random numbers table. The randomization will be done before the beginning of the study and will define which study number is going to be managed as interventional group (continuous adductor canal block - CACB) or control group (sham continuous adductor canal block - ShACB). Each patient will receive a study number following the order of their entrance on the study. The elastomeric pumps to be used connected to the catheter will be previously prepared by hospital pharmacy, accordingly to the randomization made and the subject study number, with no identification of the content (NaCl 0.9% or Ropivacaine 0.2%). Hospital pharmacy will not be blinded for which study number and elastomeric pump will be linked to the study group. Research coordinator, professional who performs the adductor canal catheter insertion and researcher who collects the data will be blinded to which group each patient was randomized. After accordance to participate on the study, the patient will be randomized to one of the two studies groups: continuous adductor canal block (CACB) or sham continuous adductor canal block (ShACB). All patients will receive the same perioperative management. The only difference will be the postoperative continuous perineural infusion: the CACB group will receive an infusion of 0.2% ropivacaine 5mL/h and ShACB group will receive an infusion of NaCl 0.9% 5mL/h. Patients will initially be brought to a dedicated block room where a safety checklist will be performed by the block room team. Standard Canadian Anesthesia Society monitoring will be provided. Mild sedation with Midazolam 0.5-2mg and Fentanyl 25-100mcg might be administered for anxiolysis and analgesia. After proper cleaning of the ipsilateral thigh, under sterile technique and ultrasound guidance (Sonosite Edge II ultrasound machine), an adductor canal block (injection of 15 mL of Ropivacaine 0.5% with epinephrine 1:200,000) and an IPACK block (injection of 15 mL of Ropivacaine 0.25% with epinephrine 1:200,000) will be performed. Cumulative local anesthetic doses will be preemptively calculated to avoid a total Ropivacaine dose of > 3mg/kg. After the peripheral nerve blocks, all patients will receive standard spinal or general anesthesia. All intraoperative opioids administered will be recorded. In the intra-operative period, each patient will receive IV Cefazolin 2g, Tranexamic acid 20mg/kg, Dexamethasone 0.1mg/kg, and Ondansetron 4mg. At the end of the procedure the surgeons will infiltrate the surgical site with 200 mg of Ropivacaine 0.2%. After surgery, the patient will be taken to the Post Anesthesia Care Unit. At this moment, an Arrow® (StimuCath® Continuous Peripheral Nerve Block Catheter) continuous adductor canal block catheter will be inserted using a Sonosite Edge II ultrasound machine. A bolus of 5-10mL of saline solution (NaCl 0.9%) with epinephrine 1:200,000 will be given, after negative aspiration, following adductor canal catheter insertion and the patient will be monitored for any heart rate change in order to rule out intravascular catheter placement. The catheter will be well secured with an adhesive fixation device to avoid displacement. Following catheter placement, the catheter will be aspirated to check for blood to ensure there is no intravascular placement.

The catheter will be aspirated prior to any injection including at the time of saline injection during catheter placement. The peripheral nerve catheter will be connected to a Baxter elastomeric pump. Depending on which group the patient is randomized to, the solution will be Ropivacaine 0.2% or Saline 0.9%. Infusion rate will be of 5mL/h. The patient will be discharged to home after achieving the discharge criteria, keeping the peripheral nerve catheter with the same infusion rate for the planed time. The adductor canal catheter will infuse for 60 hours. Prior to going home, patients will receive education and written information (educational pamphlet) regarding monitoring for local anesthetic systemic toxicity symptoms, possible CABC associated complications including potential transient muscle weakness, and instructions on patient removal of the catheter after 60 hours. This pamphlet will contain contact information for research team or Acute Pain Service, in case of any events, adverse effects or questions the patients may have about the peripheral nerve catheter. A phone number to contact each patient at home will collected before. Standard oral analgesic scheme will be prescribed to every patient (Acetaminophen 650mg QID, Celecoxib 200mg BID, Hydromorphone 1-2mg PRN Q4Hs).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary TKA in an outpatient or short-stay setting (estimated discharge on POD#0-1).
* Patients older than 21 years of age.
* American Society of Anesthesiologists (ASA) physical status I-III.
* No alcohol or drug dependency.
* Sufficient understand and co-operation about the perineural catheter.

Exclusion Criteria:

* Chronic opioid use of morphine 30mg equivalent per day for last 2 consecutive weeks.
* Allergy to the study medications.
* Coagulopathy and platelet count < 105/μL.
* Patients with contraindications to the insertion of an epidural or adductor canal catheter (severe anatomic abnormalities or history of previous surgery at the site of catheter placement).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery 15 score (QoR-15) | Day 1
  Quality of Recovery 15 score (QoR-15): from 0 to 150. Higher scores mean a better outcome.
Quality of Recovery 15 score (QoR-15) | Day 2
  Quality of Recovery 15 score (QoR-15): from 0 to 150. Higher scores mean a better outcome.
Quality of Recovery 15 score (QoR-15) | Day 3
  Quality of Recovery 15 score (QoR-15): from 0 to 150. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Pain scores | Day 1
  Numerical Rating Scale for pain (0=no pain at all; 10=worst pain)
Pain scores | Day 2
  Numerical Rating Scale for pain (0=no pain at all; 10=worst pain)
Pain scores | Day 3
  Numerical Rating Scale for pain (0=no pain at all; 10=worst pain)
Pain scores | Day 30
  Numerical Rating Scale for pain (0=no pain at all; 10=worst pain)
Opioid usage | Day 1
  Daily opioid usage in oral morphine equivalent doses
Opioid usage | Day 2
  Daily opioid usage in oral morphine equivalent doses
Opioid usage | Day 3
  Daily opioid usage in oral morphine equivalent doses
Opioid usage | Day 30
  Daily opioid usage in oral morphine equivalent doses
Catheter associated complications | Days 1, 2 and 3
  IPSILATERAL LOWER LIMB WEAKNESS; FALL; INFECTION SIGNS (REDNESS, PURULENT SECRETION, LOCAL HYPERTHERMIA) AROUND CATHETER INSERTION SITE; PRURITUS SENSATION ON INTERNAL PART OF LEG AND ANKLE; BURNING SENSATION ON INTERNAL PART OF LEG AND ANKLE; TINGLING SENSATION ON INTERNAL PART OF LEG AND ANKLE; SHOCK SENSATION ON INTERNAL PART OF LEG AND ANKLE; SIGNS OF LOCAL ANESTHETIC SYSTEMIC TOXICITY; LEAKAGE; DISCONECTION; DISLODGEMENTS / EXTERIORIZATION

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Siddiqui, MD, MSc, Principal Investigator — University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Price AJ, Alvand A, Troelsen A, Katz JN, Hooper G, Gray A, Carr A, Beard D. Knee replacement. Lancet. 2018 Nov 3;392(10158):1672-1682. doi: 10.1016/S0140-6736(18)32344-4. PMID 30496082
- [Background] Cullom C, Weed JT. Anesthetic and Analgesic Management for Outpatient Knee Arthroplasty. Curr Pain Headache Rep. 2017 May;21(5):23. doi: 10.1007/s11916-017-0623-y. PMID 28283810
- [Background] Ilfeld BM, Duke KB, Donohue MC. The association between lower extremity continuous peripheral nerve blocks and patient falls after knee and hip arthroplasty. Anesth Analg. 2010 Dec;111(6):1552-4. doi: 10.1213/ANE.0b013e3181fb9507. Epub 2010 Oct 1. PMID 20889937
- [Background] Sharma S, Iorio R, Specht LM, Davies-Lepie S, Healy WL. Complications of femoral nerve block for total knee arthroplasty. Clin Orthop Relat Res. 2010 Jan;468(1):135-40. doi: 10.1007/s11999-009-1025-1. Epub 2009 Aug 13. PMID 19680735
- [Background] Sankineani SR, Reddy ARC, Eachempati KK, Jangale A, Gurava Reddy AV. Comparison of adductor canal block and IPACK block (interspace between the popliteal artery and the capsule of the posterior knee) with adductor canal block alone after total knee arthroplasty: a prospective control trial on pain and knee function in immediate postoperative period. Eur J Orthop Surg Traumatol. 2018 Oct;28(7):1391-1395. doi: 10.1007/s00590-018-2218-7. Epub 2018 May 2. PMID 29721648
- [Background] Leung P, Dickerson DM, Denduluri SK, Mohammed MK, Lu M, Anitescu M, Luu HH. Postoperative continuous adductor canal block for total knee arthroplasty improves pain and functional recovery: A randomized controlled clinical trial. J Clin Anesth. 2018 Sep;49:46-52. doi: 10.1016/j.jclinane.2018.06.004. Epub 2018 Jun 8. PMID 29890381
- [Background] Yu R, Wang H, Zhuo Y, Liu D, Wu C, Zhang Y. Continuous adductor canal block provides better performance after total knee arthroplasty compared with the single-shot adductor canal block?: An updated meta-analysis of randomized controlled trials. Medicine (Baltimore). 2020 Oct 23;99(43):e22762. doi: 10.1097/MD.0000000000022762. PMID 33120783
- [Background] Hanson NA, Lee PH, Yuan SC, Choi DS, Allen CJ, Auyong DB. Continuous ambulatory adductor canal catheters for patients undergoing knee arthroplasty surgery. J Clin Anesth. 2016 Dec;35:190-194. doi: 10.1016/j.jclinane.2016.07.022. Epub 2016 Aug 30. PMID 27871518
- [Background] Myles PS. More than just morbidity and mortality - quality of recovery and long-term functional recovery after surgery. Anaesthesia. 2020 Jan;75 Suppl 1:e143-e150. doi: 10.1111/anae.14786. PMID 31903564
- [Background] Sun C, Zhang X, Song F, Zhao Z, Du R, Wu S, Ma Q, Cai X. Is continuous catheter adductor canal block better than single-shot canal adductor canal block in primary total knee arthroplasty?: A GRADE analysis of the evidence through a systematic review and meta-analysis. Medicine (Baltimore). 2020 May;99(20):e20320. doi: 10.1097/MD.0000000000020320. PMID 32443383
- [Background] Johansson Stark A, Charalambous A, Istomina N, Salantera S, Sigurdardottir AK, Sourtzi P, Valkeapaa K, Zabalegui A, Bachrach-Lindstrom M. The quality of recovery on discharge from hospital, a comparison between patients undergoing hip and knee replacement - a European study. J Clin Nurs. 2016 Sep;25(17-18):2489-501. doi: 10.1111/jocn.13278. Epub 2016 Jun 6. PMID 27264877